CLINICAL TRIAL: NCT02493075
Title: Ablation of Paroxysmal Atrial Fibrillation Using the Appropriate Contact Force in a Chinese Population: A Prospective Randomized Single-center Trial
Brief Title: Ablation of Paroxysmal Atrial Fibrillation Using the Appropriate Contact Force in a Chinese Population
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Chenyang Jiang, chief physician, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IIs-304
Record Dates: First submitted 2015-06-25; First posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; Catheter Ablation; contact force; Chinese-specific
MeSH Terms: conditions — Atrial Fibrillation | interventions — Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CF guided group (Experimental): Ablation will be performed with smart-touch catheter.The operator will kown the real-time contact force (CF), ablation time, FTI, etc during the procedure.
  Interventions: Behavioral: The operator blinded to the contact force data or not.
- Usual ablation group (Active Comparator): Although we use the same catheter,operator will be blinded to CF data during the procedure.
  Interventions: Behavioral: The operator blinded to the contact force data or not.

INTERVENTIONS:
Behavioral: The operator blinded to the contact force data or not. — CF guided group: ablation will be performed with the guidance of real-time CF, ablation time, FTI, etc. CF will be controlled in the range of "appropriate CF", which has been defined in phase I. Circumferential PV ablation will be performed orderly, "isolated segment"," acute reconnected segment ", and "unisolated segment" will be also identified as described in phase I.
  Usual ablation group:
  Operator will be blinded to CF data, the procedure performance is the same as described in phase I.

SUMMARY:
The objective of the study is:Phase I: To validate or otherwise determine the Chinese-specific appropriate contact force during PVI in PAF.Phase II: To evaluate the effectiveness and safety of ablation guided by the appropriate contact force.

DETAILED DESCRIPTION:
Background： Atrial fibrillation (AF) is a major cause of substantial mortality and morbidity from thromboembolism, heart failure (HF), and cognitive dysfunction. With the aging of the population and improved survival after myocardial infarction and HF, AF is emerging as a major public health concern.

Recently, significant progress has been made in treatment of AF with catheter ablation, emerging as an increasingly important technique. According to the current guidelines, catheter ablation can be considered as the first-line treatment of choice for patients with drug refractory paroxysmal AF (PAF). Circumferential PV isolation (CPVI) is a widely accepted cornerstone of this procedure, but limited by an unacceptable recurrence rate, mainly due to recovery of pulmonary vein (PV) conduction.

Durable, continuous, transmural isolation of PV is one of the most important goals of radiofrequency catheter ablation (RFCA) for PAF. The contact force (CF) between the ablation catheter and target tissue was considered closely related to the ablation effectiveness. Appropriate CF should be able to generate enough tissue lesions, and avoid the complications, such as cardiac perforation, atrial-esophageal fistula. Nowadays, irrigated ablation catheters are widely used, but the CF is mostly dependent on operators' experience and feeling, unable to be precisely measured. The tissue lesion produced would be variable in different operators, and the learning curve would be time consuming.

The newly approved CF catheter enables measurement of catheter tip contact force and force vector, providing the real-time CF during ablation. It would be helpful, not only for effective lesions formation, but also for the prevention from complications.

Studies from Western-population indicated that higher long-term successful rate could be achieved by using CF catheter, and CF between 10 to 20g was adopted in most centers. It would be important to find the appropriate range of CF for Chinese populations, because of various factors including for instance thinner and smaller atrial chambers among Chinese.

Objectives Phase I: To validate or otherwise determine the Chinese-specific appropriate CF during PVI in PAF.

Phase II: To evaluate the effectiveness and safety of ablation guided by the appropriate CF Trial design and Treatment of Subjects Phase I Instrument: CARTO™, Biosense Webster, Electrophysiology（EP）recording system, Thermocool® SmartTouch™ Catheter，Lasso/Navi-Lasso catheter, etc.

NO. of cases: 20 Study duration: 2 months Strategy：Circumferential pulmonary vein isolation Procedure： Local anaesthesia, Sedation Catheters are advanced through the right/left femoral vein. After double transseptal punctures, 8F or 8.5F SL1 Swartz sheath and Steerable sheath (e.g. Agilis, St Jude) will be placed in left atrium (LA), followed by PVs' venography Establishment of the anatomical model of LA and all PVs: Respiratory gating, Point-by-Point or Fast Anatomical Mapping (FAM). When using Point-by-Point, CF would be controlled between 5 to 10g. When using FAM, the model around PVs would be adjusted by SmartTouch catheter with CF 5-10g.

Parameter setting: Power-anterior wall 35W, posterior wall 30W; Irrigated flow rate = 17-30ml/min；Impendence - up to 170Ω； Operator: Dr. Chenyang Jiang Ablation catheter could be moved if, electrical activity amplitude decrease >80%, impedance decrease >10Ω, or ablation time more than 20s.

Endpoint: Bi-directional block between left atrial and pulmonary vein (LA-PV), and no capture along CPVI line.

The operator will be blinded to CF data, which would be monitored by the assistant. When the CF is higher than 40g, the operator will be warned.

Parameters: total procedure time, model reconstruction time, power, ablation time, impedance, CF, force-time integral (FTI).

Introduction for PV ablation:

Perform circumferential PV ablation in the order.

1. When PV is isolated after circular linear ablation without touch-up ablation, 30min waiting time + isoproterenol（ISP）/adenosine triphosphate（ATP） induction would be performed to detect the acute reconnection. If there's no reconnection, each segment will be identified as "isolated segment", and the ablation CF, time, FTI, and the power of each segment will be recorded.
2. When PV isolated initially, but reconnected by 30min+ISP/ATP observation, re-isolation would be performed, and the segment with conduction gaps(GAP) will be identified as "acute reconnected segment(s)".
3. If PV isolation not achieved by initial circumferential ablation, additional ablation along the circular lesion will be performed until PV isolated, and the segment(s) re-ablated will be identified as "unisolated segment(s)", record the parameters. 30min+ISP/ATP detection will be performed after isolation, "isolated segment(s)" and "acute reconnected segment(s)" will be identified, as described above in a. and b. If the "acute reconnected segment(s)" is the same segment(s) as "unisolated segment(s)", classify to the latter group.

Analysis for appropriate CF For each segment, single variable and multiple regression analysis will be performed between the three groups ("isolated segment"," acute reconnected segment ", and "unisolated segment"), to define an "appropriate CF". The sensitivity and specificity of the "appropriate CF" will be analyzed.

Phase II:

Instrument: CARTO™, Biosense Webster, EP recording system, Thermocool® SmartTouch™ Catheter，Lasso/Navi-Lasso catheter, etc.

NO. of cases: 120 Study duration: enrollment - 12 months, follow-up - 12 months, Data analysis and papers preparation - 3 months.

Strategy：Circumferential pulmonary vein isolation Patients will be randomized with 1:1 ratio into one of the two following groups: "CF guided group" and "usual ablation group".

Procedure： The preparation, including anaesthesia, sedation, vascular access, transseptal puncture, is the same as described in phase I.

CF guided group:

After the establishment of the anatomical model of LA and all PVs (the same as phase I), ablation will be performed with the guidance of real-time CF, ablation time, FTI, etc. CF will be controlled in the range of "appropriate CF", which has been defined in phase I. Circumferential PV ablation will be performed orderly, "isolated segment"," acute reconnected segment ", and "unisolated segment" will be also identified as described in phase I.

Endpoint: bi-directional block between LA-PV, and no capture along CPVI line. Parameters recording: total procedure time, model reconstruction time, power, ablation time, impedance, CF, FTI.

Usual ablation group:

Operator will be blinded to CF data, the procedure performance is the same as described in phase I.

Follow-up Warfarin or new oral anticoagulants will be administered to all patients for at least 3months after the procedure. The international normalized ratio will be controlled between 2.0 and 3.0 if warfarin prescribed.

After discharge, patients will be followed up at 1, 3, 6, 9, 12months post ablation. Patients' experiences, 12-lead electrocardiograms (ECGs) and Holter monitoring (non-required at 1, 9 months) will be recorded to evaluate recurrence at each appointment (not including 1 and 3 month visit post procedure) and any visits when the patient experience symptoms that suggestive of arrhythmia. The first 3 months is considered as a blanking period.

Recurrence is defined as AF/flutter/tachycardia, lasting longer than 30s, that documented by an ECG or Holter recording, or highly suggestive symptoms, after 3 months post-procedure.

Primary end point: Freedom from AF recurrence on the ECGs and Holter monitoring at each visit during the period from 3 months to 1 years after procedure, independent of antiarrhythmic drug(AAD) therapy.

Secondary end points: (1) Freedom from AF recurrence, dependent of AAD therapy; (2)Freedom of arrhythmia-related symptoms; (3)Safety Outcomes, contain mortality (death overall and procedure-related), vascular access complications (bleeding, hematoma, pseudoaneurysm, arteriovenous fistula), periprocedural events (stroke, transient ischemic attack, cardiac tamponade, pulmonary embolism, deep vein thrombosis, other embolism, LA-esophageal fistula, Other fistula, pericardial effusion, PV stenosis, atrioventricular block, heart failure exacerbation, need for a pacemaker, phrenic nerve injury, acute coronary artery occlusion, valve injury).

Follow-up will terminate after a maximum follow-up period of 12 months. Data Management Requirements for investigators on data entry The investigator ensures that data are entered into the medical records and the Case Report Forms (CRFs) truthfully, precisely, completely, timely and legally.

Information on all patients who signed the Informed Consent Form and enter the trial when considered eligible through screening should be closely observed and recorded in the CRFs without any field left blank or missing.

All data on the CRFs should be checked against the source records for consistency.

As source documents, the CRFs should be revised only by drawing a single line with the investigator's signature and date of revision added.

Source laboratory test reports (or their copies) should be adhered to the field for adhering laboratory test reports in the medical records.

Data that are significantly high or low or outside the clinically acceptable range should be carefully verified and reviewed, and necessary explanations should be given by the investigator.

Requirements for monitors on data monitoring The monitors should pay regular visits to the sites to examine the status of signing of informed consent, screening and enrollment.

Ensure that all the CRFs are correctly filled out and are consistent with the source data.

Ensure that all the errors or missing data have been corrected or explained, and have been signed and dated by the investigator.

Changes in treatment, concomitant medications, intercurrent conditions and ECG recording should be confirmed and recorded for each subject.

Discontinuations and loss-to-follow-ups of each subject should be indicated in the CRFs.

Confirm that all the adverse events (AEs) have been filed. Establishment of database and data entry Establishment of database：A study-specific database system will be established as per the items on the CRF.

Data entry: Data will be entered concurrently by data managers through double entry.

Data review: Each data item should be verified and the discrepancies be reported. The source forms should be verified on an item-by-item basis and the errors be corrected.

In case of any doubt during data entry, the data manager may fill out a Data Query Form which will be returned to the monitor. When the investigator has resolved in writing the queries in the query form and signed, the form will be sent back to the data managers. Data Query Forms should be appropriately stored.Selection and withdrawal of subjects

Statistical analysis Phase I For each segment, single variable and multiple regression analysis will be performed between the three groups ("isolated segment"," acute reconnected segment ", and "unisolated segment"), to define an "appropriate CF". The sensitivity and specificity of the "appropriate CF" will be analyzed.

Phase II Log-rank test will be used for inter-group comparison of recurrence. Kaplan-Meier method will be used for the estimation of currency curves for all points. When considering the central effects and the important prognostic factors, Cox proportional risk model will be used to estimate the risks compared with blank with the confidence intervals.

More data for "initially-isolated segment", "initially- nonisolated segment", and "additionally-isolated segment" will be collected, and the "appropriated CF" will be re-analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 75 years
* Symptomatic PAF refractory to at least one antiarrhythmic drug
* Minimum of two episodes of recurrent self-terminating AF within prior 12 months and with latest documented episode within 6 months prior ablation procedure
* First catheter ablation
* Patient is able and willing to provide written informed consent.

Exclusion Criteria:

* Persistent or long-standing persistent AF
* >4 cardioversions in prior 12 months
* Myocardial infarction(MI), coronary artery bypass grafting(CABG) or percutaneous coronary intervention (PCI) within preceding 3 months
* Left atrial diameter >5.0 cm or <3.5 cm
* Left ventricular ejection fraction by echocardiography <40%
* New York Heart Association（NYHA）class III or IV
* History of heart surgery or any previous ablation for AF
* Intracardiac thrombus
* Females who are pregnant or breast feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation (AF) recurrence rate | one year
  Patients will be followed up at 1, 3, 6, 9, 12months post ablation. Patients' experiences, 12-lead electrocardiograms (ECGs) and Holter monitoring (non-required at 1, 9 months) will be recorded to evaluate recurrence at each appointment (not including 1 and 3 month visit post procedure) and any visits when the patient experience symptoms that suggestive of arrhythmia. The first 3 months is considered as a blanking period.Recurrence is defined as AF/flutter/tachycardia, lasting longer than 30s, that documented by an ECG or Holter recording, or highly suggestive symptoms, after 3 months post-procedure.

SECONDARY OUTCOMES:
Time Data related with procedure | intraoperative
  Total procedure time, model reconstruction time, ablation time.
Number of participants with Mortality and complications | one year
  Safety Outcomes, contain mortality (death overall and procedure-related), vascular access complications (bleeding, hematoma, pseudoaneurysm, arteriovenous fistula), periprocedural events (stroke,cardiac tamponade, pulmonary embolism, deep vein thrombosis, other embolism, LA-esophageal fistula, Other fistula, pericardial effusion, PV stenosis, atrioventricular block, heart failure exacerbation, need for a pacemaker, phrenic nerve injury, acute coronary artery occlusion, valve injury).

CONTACTS AND LOCATIONS:
Overall Officials: Chenyang Jiang, MD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China